CLINICAL TRIAL: NCT00464035
Title: The Effect of Calcium on Postprandial Lipid Profile and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); The Danish Dairy Research Foundation, Denmark (Other); FOOD Graduate School, the Royal Veterinary & Agricultural University, Denmark (Other); Danish Research Agency (Other); Dutch Dairy Organization (NZO) (Other); Pharna Vinci, Denmark (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KF 01-144/02
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Obesity
Keywords: Obesity; Calcium; Fat absorption; Postprandial lipid profile; appetite
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: high calcium intake

SUMMARY:
The purpose of this study is to investigate the effect of calcium on postprandial lipid profile and appetite.

DETAILED DESCRIPTION:
Several reports have found inverse associations between calcium intake and body weight. Intervention studies have shown that a high calcium diet resulted in a greater body weight loss than a low calcium diet. In addition, it seems that calcium from dairy products have a more profound effect than calcium from supplements. The mechanism of this additional dairy effect is not yet clear, but one possible explanation could be reduced absorption of fat in the gut. The increase in fecal fat excretion on a high calcium diet could be due to the formation of calcium-fatty acid soaps in the gut.

The long term effect of a high calcium intake have been under intense investigation, but as far as we know the acute effect of a high calcium intake have not yet been examined. A study concerning the acute effects could help us understand the effect of calcium on the absorption of fat. After a meal triglyceride (TG) is packaged with cholesterol, lipoproteins and other lipids into particles called chylomicrons. Earlier studies have shown that the fatty acid pattern of chylomicron lipids postprandial was very similar to that of the ingested fat. If we assume that calcium inhibits the absorption of fat, we would expect a reduced total plasma triglyceride concentration after a calcium-rich meal.

Appetite involves many different sensations among which hunger and satiety are the most investigated. Several different hormones are involved in the regulation of appetite. Some of these hormones are known to respond to the intake or absorption of fat. If the absorption of fat is inhibited the regulation of appetite most likely will be affected. In the long term this could be important because an increased appetite probably would increase energy intake and thereby reducing the weight loss we otherwise might have accomplished by the reduced absorption of fat.

ELIGIBILITY:
Inclusion Criteria:

* healthy meals
* BMI 24-31 kg/m2
* age between 18-50 years
* hemoglobin >8 mmol/L

Exclusion Criteria:

* donation of blood 6 months before and under the study
* milk allergy, diabetes, hypertension, hyperlipidemia, cronic infectious disease
* use of dietary supplements 3 months before and under the study
* smoking
* elite athletes
* use of medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2005-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Postprandial changes in: total plasma triacylglyceride; Chylomicron triacylglyceride; Cholesterol

SECONDARY OUTCOMES:
Postprandial changes in:insulin; glucose; CCK; Ghrelin; GLP-1, appetite measured by visual analogue scales, BCAA

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Prof. Dr., Principal Investigator — Institute of Human Nutrition, the Royal Veterinary & Agricultural University, Denmark
Locations (1):
- Institute of Human Nutrition, Copenhagen, Denmark